CLINICAL TRIAL: NCT06368297
Title: The Effect of Ketone Ester Supplementation and Ketogenic Diet on Brain Plasticity in Overweight/Obese Adults: A Neurophysiological and Resting Functional Magnetic Resonance Study (rfMRI)
Brief Title: The Effect of Ketone Ester Supplementation and Ketogenic Diet on Brain Plasticity in Overweight/Obese Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BSERE22-APP007-FED
Record Dates: First submitted 2024-02-26; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity; Cognitive Change; Psychophysiologic Reaction
Keywords: Overweight; Obesity; Ketone; Neurocognition
MeSH Terms: conditions — Overweight; Obesity; Ketosis | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute effect of ketone monoester supplementation (Experimental): To investigate the acute effect of ketone monoester ingestion on brain cortical plasticity using high-frequency rTMS.
  Interventions: Dietary Supplement: Ketone Monoester Supplementation
- Effects of a 2-week ketogenic diet or ketone monoester supplementation (Experimental): To evaluate the impact of short-term ketogenic dieting and ketone monoester supplementation on brain plasticity.
  To investigate structural and functional brain adaptations to short-term ketogenic dieting and ketone supplementation.
  To assess the relationship between changes in brain plasticity and the brain's structural and functional adaptations and changes in circulating levels of brain-derived neurotrophic factors and key central acting hormones (i.e., insulin and leptin) due to ketogenic dieting and ketone monoester supplementation.
  Interventions: Dietary Supplement: Ketone Monoester Supplementation; Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketone Monoester Supplementation — Exogenous ketones are a class of ketone bodies that are ingested using nutritional supplements or foods. This class of ketone bodies refers to the three water-soluble ketones (acetoacetate, β-hydroxybutyrate [β-HB], and acetone).
Dietary Supplement: Ketogenic diet — The ketogenic diet typically reduces total carbohydrate intake to less than 50 grams a day-less than the amount found in a medium plain bagel-and can be as low as 20 grams a day. Generally, popular ketogenic resources suggest an average of 70-80% fat from total daily calories, 5-10% carbohydrate, and 10-20% protein.
  Arms: Effects of a 2-week ketogenic diet or ketone monoester supplementation

SUMMARY:
This project comprises an initial crossover placebo-controlled neurophysiological study to ascertain the effect of acute ketone ester ingestion on motor cortex plasticity, followed by a second 2-week intervention study aimed to compare the effect of a ketogenic diet versus ketone ester supplementation on motor cortex plasticity, resting brain function and structure, and metabolic and neuroendocrine responses.

DETAILED DESCRIPTION:
The study initially makes a bold attempt to explore whether the ketone supplementation would induce improvements in the overweight/ obese population's brain health via altering motor cortex plasticity, brain function and structure, and metabolic and neuroendocrine pathways. The study's aims include:

* assessing changes in brain plasticity associated with excessive body weight and/or obesity.
* evaluating the potential of ketone monoester supplementation in enhancing brain plasticity.
* evaluating the potential of ketone monoester supplementation in correcting impaired brain plasticity due to excessive body weight.
* evaluating the impact of short-term ketogenic dieting and ketone monoester supplementation on brain plasticity.
* investigating structural and functional brain adaptations to short-term ketogenic dieting and ketone supplementation.
* assessing the relationship between changes in brain plasticity and the brain's structural and functional adaptations and changes in circulating levels of brain-derived neurotrophic factors and key central acting hormones (i.e., insulin and leptin) due to ketogenic dieting and ketone monoester supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 25 and < 35 kg/m2 (overweight/obese group) or BMI > 18.5 and < 25 kg/m2 (healthy weight group);
* Right-handed.

Exclusion Criteria:

* Presenting any established counter indication for transcranial magnetic stimulation;
* Currently taking any medication affecting the central or the peripheral nervous system;
* Suffering from any psychiatric, neurologic, cardiovascular, or metabolic disease, including type 1 and type 2 diabetes mellitus;
* Undertaking surgery in the past six months;
* Engaged in resistance training.
* Pregnancy;
* Breastfeeding;
* Being amenorrhea.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Brain Plasticity | 2 weeks
  This measurement is "brain plasticity". Brain plasticity, also known as neuroplasticity, refers to the brain's remarkable ability to change and adapt in response to experience. The brain plasticity will be measured by transcranial magnetic stimulation (TMS) system. When assessing brain plasticity using TMS through the measurement of Motor Evoked Potentials (MEPs), the primary unit of measurement is typically in millivolts (mV) for the amplitude of the MEPs. MEPs are electrical signals recorded from muscles after stimulation of the motor cortex with TMS, reflecting the excitability of the corticospinal pathway and, indirectly, cortical plasticity.
Grey Matter Volume | 2 weeks
  The measurement name is "grey matter volume", which belongs to brain structure. The grey matter volume will be assessed by the magnetic resonance imaging system. Grey matter volume is generally measured in cubic centimeters (cm³) or milliliters (mL), as both units are equivalent in volume measurement (1 cm³ = 1 mL). This measure reflects the volume of grey matter regions in the brain, which include areas dense with neuronal cell bodies, dendrites, axon terminals, and glial cells.
Cortical Thickness | 2 weeks
  The measurement name is "cortical thickness", which belongs to brain structure. The cortical thickness will be assessed by the magnetic resonance imaging system. Cortical thickness is measured in millimeters (mm). It refers to the average thickness of the grey matter cortex across various regions of the brain. Cortical thickness can vary significantly across different parts of the cortex, typically ranging from around 1 mm to 4 mm, depending on the specific brain region and individual differences.
Blood-Oxygen-Level-Dependent (BOLD) Signal Changes | 2 weeks
  The measurement name is "Blood-Oxygen-Level-Dependent (BOLD) Signal Changes", which belongs to brain function. The cortical thickness will be assessed by the magnetic resonance imaging system (MRI). The unit of BOLD signal changes measured by MRI is typically expressed as a percentage change (%). The BOLD signal reflects changes in the magnetic properties of blood due to variations in oxygenation levels that occur in response to neural activity.

SECONDARY OUTCOMES:
Blood Glucose | 6 weeks
  The measurement name is "blood glucose". It will be assessed by a glucometer in laboratory settings. The unit of measurement is millimoles per liter (mmol/L).
Blood Beta-Hydroxybutyrate | 6 weeks
  The measurement name is "blood beta-hydroxybutyrate". It will be assessed by specific ketone meters designed for beta-hydroxybutyrate measurement. The unit of measurement is millimoles per liter (mmol/L).
Blood Insulin | 6 weeks
  The measurement name is "blood insulin". It will be assessed by immunoassay system (chemiluminescence immunoassay analyzer) using blood samples. The unit of measurement is microunits per milliliter (μU/mL).
Leptin | 6 weeks
  The measurement name is "leptin". It will be assessed by immunoassay system (chemiluminescence immunoassay analyzer) using blood samples. The unit of measurement is nanograms per milliliter (ng/mL).
Ghrelin | 6 weeks
  The measurement name is "ghrelin". It will be assessed by immunoassay system (chemiluminescence immunoassay analyzer) using blood samples. The unit of measurement is picograms per milliliter (pg/mL).
Brain-Derived Neurotrophic Factor | 6 weeks
  The measurement name is "brain-derived neurotrophic factor". It will be assessed by immunoassay system (chemiluminescence immunoassay analyzer) using blood samples. The unit of measurement is nanograms per milliliter (ng/mL).
Reaction Time of Attention Network Test | 2 weeks
  The measurement name is "reaction time of Attention Network Test". The measurement will be assessed by psychological paradigm named Attention Network Test. The unit of measurement is milliseconds (ms).
Accuracy of Attention Network Test | 2 weeks
  The measurement name is "accuracy of attention network test". The measurement will be assessed by psychological paradigm named Attention Network Test. Accuracy is generally measured as a percentage (%).
Reaction Time of Stroop Task | 2 weeks
  The measurement name is "reaction time of stroop task". The measurement will be assessed by psychological paradigm named Stroop Task. The unit of measurement is milliseconds (ms).
Accuracy of Stroop Task | 2 weeks
  The measurement name is "accuracy of stroop task". The measurement will be assessed by psychological paradigm named Stroop Task. Accuracy is generally measured as a percentage (%).
Reaction Time of N-back Task | 2 weeks
  The measurement name is "reaction time of n-back task". The measurement will be assessed by psychological paradigm named N-back task. The unit of measurement is milliseconds (ms).
Accuracy of N-back Task | 2 weeks
  The measurement name is "accuracy of n-back task". The measurement will be assessed by psychological paradigm named N-back task. Accuracy is generally measured as a percentage (%).
Cerebral Hemoglobin Concentration | 2 weeks
  The measurement name is "cerebral hemoglobin concentration". The measurement will be assessed by functional near-infrared spectroscopy (fNIRS). The unit of measurement is micromoles per liter (μM).
Height in Kilograms | 2 weeks
  The measurement name is "height in kilograms". It will be assessed by a stadiometer. The unit of measurement is meters (m).
Weight in Meters | 2 weeks
  The measurement name is "weight in meters". It will be assessed by a scale. The unit of measurement is kilograms (kg).
Body Fat Percentage | 2 weeks
  The measurement name is "body fat percentage". It will be assessed by a bioelectrical impedance analysis device. The unit of measurement is percentage (%).
Fat Mass | 2 weeks
  The measurement name is "fat mass". It will be assessed by a bioelectrical impedance analysis device. The unit of measurement is kilograms (kg).
Muscle Mass | 2 weeks
  The measurement name is "muscle mass". It will be assessed by a bioelectrical impedance analysis device. The unit of measurement is kilograms (kg).
Body Water | 2 weeks
  The measurement name is "body water". It will be assessed by a bioelectrical impedance analysis device. The unit of measurement is liters (L).
Body Mass Index | 2 weeks
  The measurement name is "body mass index (BMI)". It will be assessed by calculating BMI using height and weight measurements obtained from a stadiometer and a scale, respectively. The unit of measurement is kilograms per square meter (kg/m²).
Skinfold Thickness | 2 weeks
  The measurement name is "skinfold thickness". It will be assessed by skinfold calipers. The unit of measurement is millimeters (mm).
Maximal Oxygen Uptake | 2 weeks
  The measurement name is "maximal oxygen uptake". It will be assessed by cardiopulmonary exercise testing (CPET) equipment, such as cycle ergometers, along with a metabolic cart for measuring oxygen consumption. The unit of measurement is milliliters of oxygen per kilogram per minute (mL/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: Zhaowei Kong, PhD, Principal Investigator — University of Macau

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared by request two years after the completion. The data will be available for two years.
Supporting Information: Study Protocol, SAP
Time Frame: 01/09/2026-01/09/2028
Access Criteria: The data will be shared by request two years after the completion. The data will be available for two years.

REFERENCES:
- [Background] Falkenhain K, Daraei A, Forbes SC, Little JP. Effects of Exogenous Ketone Supplementation on Blood Glucose: A Systematic Review and Meta-analysis. Adv Nutr. 2022 Oct 2;13(5):1697-1714. doi: 10.1093/advances/nmac036. PMID 35380602
- [Background] Evans M, McClure TS, Koutnik AP, Egan B. Exogenous Ketone Supplements in Athletic Contexts: Past, Present, and Future. Sports Med. 2022 Dec;52(Suppl 1):25-67. doi: 10.1007/s40279-022-01756-2. Epub 2022 Oct 10. PMID 36214993
- [Result] Kesl SL, Poff AM, Ward NP, Fiorelli TN, Ari C, Van Putten AJ, Sherwood JW, Arnold P, D'Agostino DP. Effects of exogenous ketone supplementation on blood ketone, glucose, triglyceride, and lipoprotein levels in Sprague-Dawley rats. Nutr Metab (Lond). 2016 Feb 4;13:9. doi: 10.1186/s12986-016-0069-y. eCollection 2016. PMID 26855664
- [Result] Walsh JJ, Neudorf H, Little JP. 14-Day Ketone Supplementation Lowers Glucose and Improves Vascular Function in Obesity: A Randomized Crossover Trial. J Clin Endocrinol Metab. 2021 Mar 25;106(4):e1738-e1754. doi: 10.1210/clinem/dgaa925. PMID 33367782
- [Derived] Yu Q, Wong KK, Lei OK, Armada-da-Silva PAS, Wu Z, Nie J, Shi Q, Kong Z. Acute ketone monoester supplementation in young adults: modulating metabolic and neurocognitive functions across body weights. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-12. doi: 10.1139/apnm-2024-0229. Epub 2024 Oct 17. PMID 39418669